CLINICAL TRIAL: NCT03762356
Title: What Factors Are Important When Assessing an Individual's Insight/Awareness of Their Own Violence Risk?
Brief Title: Questionnaire About Individual's Insight/Awareness of Risk of Violence
Status: Withdrawn | Type: Observational
Why Stopped: Study did not receive final approval however it was decided to not pursue.
Sponsor: Bournemouth University (Other)
Collaborators: Dorset HealthCare University NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: BournemouthU
Record Dates: First submitted 2018-10-03; First posted 2018-12-03 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Risk Behavior, Health; Violence; Risk Behavior
Keywords: Insight; Awareness; Violence; Professional views; Risk to others
MeSH Terms: conditions — Health Risk Behaviors; Risk-Taking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall aim of this questionnaire is to gather the views of qualified clinicians on what factors contribute to an individual's insight or awareness into their own violent behaviours. The questionnaire will also explore what type of tool would be useful to develop for use in clinical practice to aid effective risk assessment and management. Brief demographic information will also be gathered.

DETAILED DESCRIPTION:
Despite insight into violence being a factor regularly addressed by professionals in the assessment of future violence occurring research on this concept is sparse. Research instead tends to focus specifically on insight into violence specifically in relation to schizophrenia rather than more broadly in forensic and other clinical settings. What evidence there is suggests that developing an individual's insight or awareness of their own risk of violence is a key factor in reducing the likelihood of them engaging in further acts of violence. Being able to appropriately assess this is key and appears to currently be inconsistent between professionals.

In this study, therefore, a questionnaire will be disseminated to professionals working in secure care or a forensic community setting in order to gather their views on what factors contribute to an individual's insight or awareness into their own violent behaviours.

All clinicians/professionals who are currently employed and qualified as an Offender Manager, Offender Supervisor, Psychologist, Nurse, Social Worker, Occupational Therapist, Psychiatrist, Prison Officer currently working in a secure care or forensic community setting will be eligible to participate. Individuals with the appropriate qualifications working within private practice in the UK will also be eligible to participate. Those working outside the UK will not be eligible to participate.

ELIGIBILITY:
Inclusion Criteria:

* Employed as a qualified as a Psychologist, Nurse, Social Worker, Occupational Therapist, Psychiatrist, Prison Officer or Offender Manager currently working in a secure care or forensic community setting.

Exclusion Criteria:

* Those working solely in private practice outside of organisations and those who work outside the UK, are not eligible to participate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Employed as a qualified as a Psychologist, Nurse, Social Worker, Occupational Therapist, Psychiatrist, Prison Officer or Offender Manager currently working in a secure care or forensic community setting
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Questionnaire responses that measure levels of insight or awareness of violence | 10 minutes
  Online survey responses as to range of factors identified by clinicians, a consensus on a format of insight tool and to have sufficient information to be able to devise an insight tool that measures level of insight or awareness of violence.

CONTACTS AND LOCATIONS:
Overall Officials: Joe Lowenstein, BSc MSc DClinPsy, Study Chair — Chief Investigator

IPD SHARING:
Plan to Share IPD: No